CLINICAL TRIAL: NCT01487642
Title: Study of the Effect of Two Different Types of Telephone Counselling Respectively and a Web-based Smoking Cessation Programme Among Adult Daily Cigarette Smokers.
Brief Title: Comparison of Four Different Smoking Cessation Programmes
Acronym: Fristart
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: Danish Cancer Society (Other); National Board of Health, Denmark (Other Government)
Responsible Party: Principal Investigator, Peter Dalum, Primary investigator, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIPH-2066
Record Dates: First submitted 2011-11-24; First posted 2011-12-07 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Smoking; Smoking Cessation; Self-efficacy
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Telephone counselling (Experimental)
  Interventions: Device: Standard 15-minute telephone counselling; Device: Proactive telephone counselling
- Proactive telephone counselling (Experimental)
  Interventions: Device: Proactive telephone counselling
- web-based smoking cessation programme (Experimental)
  Interventions: Device: Interactive web-based smoking cessation programme
- Self-help material (Active Comparator)
  Interventions: Device: Self-help material

INTERVENTIONS:
Device: Standard 15-minute telephone counselling — Subjects in arm 1 will benefit from a standard 15-minute telephone counselling session with a professional adviser which resembles a normal call to the national Quit-line. The telephone counselling will be reactive, thus the smoker initiates the call to a designated number to receive advice and information based on the needs and wishes of this particular smoker. Participants can receive self-help materials and information on other smoking cessation services if they wish.
  Other Names: Stoplinien.dk
  Arms: Telephone counselling
Device: Proactive telephone counselling — subjects in arm 2 will benefit from of five 15-minute calls from a professional adviser. Similar to the standard reactive telephone counselling, the proactive counselling will be a personal discussion and advice based on the needs and wishes of the particular participant. Together, the participant and adviser will determine a cessation date and schedule one call 3-7 days before the cessation date, one call immediately after the cessation date and three additional calls on days 3, 10 and 24, respectively, post-cessation.
  Other Names: Stoplinien.dk
  Arms: Proactive telephone counselling; Telephone counselling
Device: Interactive web-based smoking cessation programme — Subjects in arm 3 will benefit from a tailored and interactive web-based smoking cessation programme. Besides interactive and personalised information generated on the webpage, the participant will receive by e-mail and SMS tailored feedback messages based on the particular profile of the participant on particular dates as well as topics during the cessation period depending on how well the cessation is proceeding.
  Other Names: ddsp.dk
  Arms: web-based smoking cessation programme
Device: Self-help material — Participants receives self-help materials and on request information on other smoking cessation services if they wish.
  Other Names: stoplinien.dk
  Arms: Self-help material

SUMMARY:
The primary objective of the study is to compare the efficacy of four different smoking cessation programmes, including a proactive telephone counseling intervention, a reactive telephone counseling a and an interactive web-based intervention and (as control) written self-help material.

DETAILED DESCRIPTION:
Smoking remains the most important threat to public health. The majority of smokers wish to quit smoking and every year a substantial part of smokers makes a quit attempt. However, the majority of smokers tries to quit unassisted and existing smoking cessation interventions are underused. In this study we test the effectiveness of four different smoking cessation interventions in a randomized controlled trial. The study provides knowledge on factors important for recruitment and gives indication on potential reach of interventions among the general population. This knowledge can help us in designing interventions that is both effective but also have a high reach in the general population.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16 and older
* Current smoker: Willing to quit smoking within the next 12 weeks
* Having a regular access to Internet
* Having a personal e-mail address
* Having a personal mobile cell phone with a Danish number
* Given informed consent
* Can read and understand Danish

Exclusion Criteria:

* Less than 16 years of age
* No personal e-mail address
* No personal mobile cell phone
* Not able to give informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Smoking cessation | 14 months post baseline
  We measure the 30 days point prevalence abstinence rate. We measure whether participants have been totally smokefree for at least 30 days prior to the follow-up date.

SECONDARY OUTCOMES:
Smoking cessation | 3 month post baseline
  We measure the 30 days point prevalence abstinence rate. We measure whether participants have been totally smokefree for at least 30 days prior to the follow-up date.
smoking cessation | 8 month post baseline
  We measure the 30 days point prevalence abstinence rate. We measure whether participants have been totally smokefree for at least 30 days prior to the follow-up date.
Change in self-efficacy | At 3, 8 and 14 months
  Self-efficacy (SE) is measured on a 12 item scale. SE describes the individuals belief in own capacity to refrain from smoking in 12 specific situations. SE change is defined af the difference between baseline SE and SE at the 3,8 and 14 months follow-ups.
Motivational change | At 3, 8 and 14 months
  Motivation was measured on a 10 point scale. ("How important is it for you to quit smoking"). Motivational change is defined af the difference between baseline motivation and motivation at the 3,8 and 14 months follow-ups.
Stage of change | At 3, 8 and 14 months
  A measure of the participants intentions to quit smoking in the future ("Do you have plans to quit smoking? yes, within the next 30 days; yes, within the next six months; yes, but I no specific plans; No").
Smoking cessation expectations | at 3,8,14 months
  We look at differences from baseline to follow-up with regard to participants perception of being smokefree on a six item scale: activities, physical fitness, health, appearance, happiness, stress.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Dalum, Ph.d, Principal Investigator — University of Southern Denmark
Locations (1):
- National institute of Public Health, University of Southern Denmark, Copenhagen, Denmark

REFERENCES:
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Skov-Ettrup LS, Dalum P, Bech M, Tolstrup JS. The effectiveness of telephone counselling and internet- and text-message-based support for smoking cessation: results from a randomized controlled trial. Addiction. 2016 Jul;111(7):1257-66. doi: 10.1111/add.13302. Epub 2016 Apr 13. PMID 26748541